CLINICAL TRIAL: NCT05098561
Title: Music Therapy as a Supplement to Post Surgery Pain Management in Cardiac Surgery Patient Following Median Sternotomy
Brief Title: Music Therapy for Post-cardiac Surgery Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Principal Investigator, Stanley Tam, Attending Surgeon, Steward St. Elizabeth's Medical Center of Boston, Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00770
Record Dates: First submitted 2021-09-18; First posted 2021-10-28 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Opioid Use

STUDY DESIGN:
Intervention Model Description: Randomize patients into music treatment group and non-music treatment control group. 30 patients per group. Patients will be enrolled into each group on an alternate bases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music treatment group (Experimental): The nurse will set up the appropriate music genre for the each music treatment patient, based on patient's preference obtained from the pre-operative questionnaire, by using the bedside computer and using Pandora, the internet music streaming service.
  Interventions: Other: Music Treatment
- Control Group (No Intervention): No music treatment will be used. Standard pain and comfort measure only.

INTERVENTIONS:
Other: Music Treatment — The nurse will set up the appropriate music genre for the each music treatment patient, based on patient's preference obtained from the pre-operative questionnaire, by using the bedside computer and using Pandora, the internet music streaming service.
  Arms: Music treatment group

SUMMARY:
Music therapy as a supplement to post surgery pain management in cardiac surgery patients following median sternotomy.

DETAILED DESCRIPTION:
2. Specific Aims:

1. Primary Aim: To assess whether music therapy can decrease the amount of opioid type pain medications used.

   Hypothesis: Music therapy reduces the amount of opioid type pain medication used in management of post-operative pain and discomfort.
2. Secondary Aims:

i. To identify the gender and age groups of patients who can benefit from music therapy as a supplement to post-operative pain management.

Hypothesis: Majority of the population of patient benefits from music therapy as a supplement to postoperative pain management.

ii. To assess whether music therapy can increase patient satisfaction.

Hypothesis: Music therapy increases patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery via median sternotomy

Exclusion Criteria:

* Emergency cases.
* Patients with hearing impairment.
* Patients with dementia or other mental status changes.
* Patients who are clinically unstable postoperatively.
* Patients who develop postoperative complications.
* Patients who are non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-09-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
The amount of Opioid type pain medication used | In the immediate post operative period, while patient still in the ICU
  To assess whether the use of music therapy can decrease the amount of opioid type pain medications used.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Tam, Principal Investigator — Steward St Elizabeth Medical Center
Locations (1):
- Steward St. Elizabeth medical Center, Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No